CLINICAL TRIAL: NCT02839512
Title: A Trial of the Jejunal to Ileal Diversion Endoscopic Procedure (Side-to-Side Anastomosis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIW 14-001
Record Dates: First submitted 2016-07-11; First posted 2016-07-21 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Jejunal to Ileal Diversion (Experimental): All subjects who receive jejunal to ileal diversion endoscopic procedure
  Interventions: Device: Jejunal to Ileal Diversion

INTERVENTIONS:
Device: Jejunal to Ileal Diversion — The Jejunal to Ileal Diversion procedure will be performed using colonoscopes to place magnets to create a side to side compression anastomosis. The colonoscope delivered magnet creates the proximal end of the anastomosis approximately 100 cm distal from the ligament of Treitz. The colonoscope delivered magnets creates the distal end of the anastomosis approximately 100 cm proximal from the ileocecal junction.

SUMMARY:
This is a single center study to assess metabolic effects in subjects after a Jejunal to Ileal Diversion procedure was performed using colonoscopes.

DETAILED DESCRIPTION:
The Jejunal to Ileal Diversion procedure is an adaptation of a biliopancreatic diversion with duodenal switch, which is a surgical procedure used to treat metabolic syndrome conditions. The small bowel diversion of the jejunum into the ileum by creating a single anastomosis just beyond the ligament of Trietz will be studied. Up to 15 eligible subjects will be enrolled into the trial. Enrollment will stop once 10 subjects have undergone the Jejunal to Ileal Diversion procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* A BMI ≥ 30 kg/m2 and < 50 kg/m2 If subject has Type 2 Diabetes
* HbA1c ≥ 6.5% and ≤ 9%
* Fasting plasma glucose greater than 110 mg/dl
* Treatment with up to 2 oral diabetic medications
* Able to understand and sign informed consent document
* If subject is female, she must commit to not becoming pregnant for 18 months and agree to use of contraceptives during this period

Exclusion Criteria:

* Any conditions for which endoscopy/colonoscopy would be contraindicated.
* Congenital or acquired anomalies of the GI tract, including atresias, stenosis or malrotation.
* Previous abdomino-pelvic surgery that may result in adhesions or anatomical changes that may interfere with placement of the GIW device.
* Diagnosis of Type 2 diabetes less than 6 months
* More than 2 oral diabetic medications
* Use of insulin
* If on metformin, history of polycystic ovarian syndrome (PCOS)
* Use of Dipeptidyl peptidase-4 (DPP-4) inhibitors
* Use of GLP-1 agonists
* Use of Use of alpha-glucosidase inhibitors
* Type 1 Diabetes
* Unable or unwilling to perform home blood glucose monitoring
* History of or suspected gastrointestinal disease (e.g. cirrhosis, inflammatory bowel disease)
* History of active malignancy (i.e. not in remission) with the exception of squamous or basal cell carcinoma of the skin
* Any blood coagulation disorder
* Implanted cardiac pacemaker, defibrillator or other implanted electric device - Ongoing systemic infection
* Chronic pancreatitis
* Chronic liver disease of any cause
* Poorly controlled psychiatric disease (e.g. ongoing major depression, schizophrenia, borderline personality, suicidality, psychosis)
* Any history of an eating disorder within the past 5 years
* Pre-existing severe comorbid cardio-respiratory disease (e.g. congestive heart failure, cardiac arrhythmia, coronary artery disease, chronic obstructive lung disease, pulmonary embolism)
* Uncontrolled hypertension (systolic BP > 150 mm Hg or diastolic BP > 100 mm Hg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin A1c | 12 months
  Difference from baseline HbA1c at baseline and HbA1c at 12 months

SECONDARY OUTCOMES:
Weight loss (%TBWL) | 12 months
  Difference from baseline total body weight loss at baseline and total body weight loss at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Evžen Machytka, Principal Investigator — University of Ostrava Hospital

IPD SHARING:
Plan to Share IPD: No
12 Month Study results published in Gastrointestinal Endoscopy in 2017

REFERENCES:
- [Result] Machytka E, Buzga M, Zonca P, Lautz DB, Ryou M, Simonson DC, Thompson CC. Partial jejunal diversion using an incisionless magnetic anastomosis system: 1-year interim results in patients with obesity and diabetes. Gastrointest Endosc. 2017 Nov;86(5):904-912. doi: 10.1016/j.gie.2017.07.009. Epub 2017 Jul 14. PMID 28716404